CLINICAL TRIAL: NCT07198386
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of CS060380 Tablets in Patients With Non-alcoholic Steatohepatitis (NASH).
Brief Title: Trial of CS060380 Tablets for Non-alcoholic Steatohepatitis (NASH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS060380-NASH-CN-IIa-02
Record Dates: First submitted 2025-09-08; First posted 2025-09-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: NASH

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: 0.25 mg CS060380 (Experimental): Take five tablets of 0.05mg CS060380 daily for 12 weeks.
  Interventions: Drug: CS060380
- Group B: 0.5 mg CS060380 (Experimental): Take one tablet of 0.5mg CS060380 and four tablets of placebo daily for 12 weeks.
  Interventions: Drug: CS060380; Drug: Placebo
- Placebo (Placebo Comparator): Take five tablets of placebo daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CS060380 — Oral QD
  Arms: Group A: 0.25 mg CS060380; Group B: 0.5 mg CS060380
Drug: Placebo — Oral QD
  Arms: Group B: 0.5 mg CS060380; Placebo

SUMMARY:
The goal of this clinical trial is to learn if CS060380 tablets works to treat non-alcoholic steatohepatitis(NASH) in adults.It will also learn about the safety of CS060380 tablets.The main questions it aims to answer are:

* After 12 weeks of administration, what was the percentage change in fat content evaluated by MRI-PDFF compared to the baseline？
* What medical problems do participants have when taking CS060380 tablets? Researchers will compare CS060380 tablets to a placebo (a look-alike substance that contains no drug) to see if CS060380 tablets works to treat NASH.

Participants will:

* Take CS060380 tablets or a placebo every day for 12 weeks
* Visit the clinic for checkups and tests at the frequency required by the protocol
* Keep a diary of their symptoms and the number of tablets taken

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled Phase IIa clinical trial to evaluate CS060380 tablets in patients with non-alcoholic steatohepatitis (NASH).

Subjects who meet the inclusion criteria will be randomly assigned in a 1:1:1 ratio to study group A at 0.25mg, study group B at 0.5mg, and placebo group, with a planned inclusion of 20 subjects in each group. They will take the investigational product on an empty stomach once a day at a fixed time as much as possible for 12 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 70 (including the boundary value).
2. Liver biopsy results within 6 months prior to randomization were consistent with the pathological diagnosis of NASH, and the non-alcoholic fatty liver disease activity score (NAS) was ≥4 points, with at least 1 point each for inflammation and balloon changes, and the fibrosis stage of the Clinical Study Network for Non-alcoholic Steatohepatitis (NASH-CRN) in the United States was F1-F3; Or magnetic resonance proton density fat content measurement (MRI-PDFF) within 3 months prior to randomization confirmed that the liver fat content was ≥10%.
3. Participants with fertility and their spouses or partners voluntarily took effective contraceptive measures from screening to within 3 months after the last administration. Among them, women of childbearing age include premenopausal women and women within two years after menopause, except those who have undergone hysterectomy or bilateral oophorectomy or have medically confirmed ovarian failure.
4. Stable ALT and AST results before randomization. If the ALT or AST value during the screening period is greater than 1.5× upper limit of normal (ULN), there must be two consecutive stable evidences before randomization (with an interval of at least 2 weeks between the two evaluations), and one of the following evidences must be met:

   * Compared with the historical data within 2 weeks to 3 months before randomization (if any, and the value ≤5×ULN), the ALT or AST value during the screening period needs to increase by ≤30% compared with the historical data.
   * If there is no available historical data and the ALT or AST value during the screening period is greater than 1.5×ULN, the test should be repeated at least once every two weeks. The ALT or AST value after re-testing should increase by no more than 30% compared to the screening period.
5. Avoid strenuous exercise at least 24 hours before each visit or blood draw.
6. Sign the ICF before the experiment and be able to complete the research as required by the protocol.

Exclusion Criteria:

1. The following liver diseases or past medical history were present at the time of screening:

   1. Patients with other clinically significant acute or chronic liver diseases or biliary tract diseases not caused by NASH, and the researchers determined that not suitable to participate in this study, Including but not limited to hepatitis B virus, Untreated hepatitis C virus, DILI, ALD, WD, AIH, PBC, PSC.
   2. Has a history of liver cirrhosis.
   3. Primary liver cancer. AFP > 50 μg/L.
2. During screening, the following medical history was present:

   1. Study the history of allergies to drug ingredients and excipients.
   2. Surgical procedures that may interfere with treatment, including but not limited to weight loss surgery, liver transplantation surgery, etc.
   3. Screen those who have a history of malignant tumors within the previous five years.
   4. Contraindications for any MRI scan.
   5. Screen for a history of drug or substance abuse within the previous two years.
   6. Screen for a history of heavy drinking for more than three consecutive months within one year prior to the screening.
   7. Weight change ≥ 5% in the first 3 months of randomization or ≥ 10% in the first 6 months of randomization.
   8. Individuals who have donated blood within the past 3 months prior to screening, and those who have lost a total of 400 mL or more due to blood donation or other reasons within the past 6 months.
   9. Merge with any of the following serious cardiovascular disease or surgical histories (including but not limited to):

      1. Unstable angina pectoris occurred within 3 months prior to randomization.
      2. Combined heart failure, NYHA ≥ Ⅲ
      3. Myocardial infarction, shock or life-threatening arrhythmia occurred within 6 months prior to randomization.
      4. Randomized coronary artery bypass grafting surgery or percutaneous coronary intervention within the first 6 months.
3. The following concomitant diseases or conditions occur during the screening period:

   1. T1DM, uncontrolled T2DM (HbA1c > 9 % ), history of severe hypoglycemia.
   2. Intestinal diseases that affect the absorption of oral medications.
   3. There are thyroid diseases, including hyperthyroidism and hypothyroidism or pituitary disorders.
   4. Combined with serious diseases such as circulatory, respiratory, urinary, hematological, immune, psychiatric, neurological, and renal disorders, it has been determined by the researchers that it is not suitable to participate in this study.
   5. Uncontrolled hypertension was present during screening: systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg even under regular medication control.
   6. When screening QTcF >450 ms (for males) or >470 ms (Female).
   7. When screening, HIV antibody positive and syphilis spiral antibody positive.
   8. Pregnant and lactating women.
   9. Laboratory test:

      1. PLT<LLN.
      2. TBIL > 1.2×ULN, Gilbert Syndrome.
      3. ALT or AST > 5 × ULN.
      4. eGFR < 50 mL/min/1.73 m².
      5. IRN > 1.5.
      6. THS or FT4 abnormality.
      7. Cardiac Troponin > ULN.
4. The following medication history existed before randomization:

   1. No stable dose of sodium-glucose cotransporter-2 was received within 6 months prior to randomization(SGLT2).
   2. Use of an excessively high dose of vitamin E within 6 months prior to randomization (unless the dose is stable and <400 IU/d), pioglitazone, glucagon-like peptide-1 (GLP-1) receptor agonists GIPR/GLP-1R dual agonists, GIPR/GLP-1R/GCGR triple agonists, compound Oral antidiabetic (OAD) regimens (three or more OADs).
   3. Those who have received treatment for NAFLD/NASH including but not limited to the following within 3 months prior to randomization Drugs, FXR agonists, FGF21 analogues, DGAT2 inhibitors, PDE inhibitors Agents, other THR-β agonists, obeticholic acid, etc.
   4. Within 3 months prior to randomization (for unmarketed drugs or devices) or within 5 half-lives (for marketed drugs), the patient has participated in other investigational product or device clinical trials (if there is evidence that the patient participated in a clinical trial, received treatment in the inactive drug group, or has been removed from the group without receiving treatment with the investigational product, they are eligible to participate in this study for screening).
   5. Having received drug treatment that includes but is not limited to the following drugs that may cause NAFLD/NASH for at least 2 weeks within one month prior to boarding the machine For example, total parenteral nutrition (TPN), amiodarone, methotrexate, systemic glucocorticoids, tetracycline, tamoxifen, estrogen with doses greater than those used for contraception or hormone replacement, anabolic steroids, valproic acid and other known liver-toxic drugs.
   6. Within 4 weeks prior to randomization or during the intended clinical study period, liver-protecting drugs not permitted by the protocol were used, including but not limited to silymarin (bin), bicyclol, glycyrrhizic acid preparations (magnesium isoglycyrrhizinate, compound glycyrrhizin, diammonium glycyrrhizinate, etc.).
   7. Received anticoagulant treatment within 2 weeks prior to randomization: drugs that increase INR (e.g., FXa inhibitors, warfarin, heparin, etc.).
   8. Those who have used CYP3A enzyme strong suppressors, CYP3A enzyme strong inducers, inhibitors of P-gp or BCRP transporters that may affect the metabolism or absorption of this drug within 14 days prior to randomization or at least 5 half-lives (whichever is longer).
5. Other circumstances that the researcher deems unsuitable for inclusion in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
MRI-PDFF | D85
  To assess the changes in liver steatosis through magnetic resonance imaging (MRI) proton density fat fraction (PDFF) from baseline to Week 12.

SECONDARY OUTCOMES:
AE, SAE, Vital signs, Physical examination, 12-ECG, Thyroid function, laboratory tests. | Up to 12 weeks
  Safety and Tolerability.
ALT, AST, GGT, TC, LDL-C, HDL-C, TG, ApoB, Lp(a), VLDL, The ApoB/ApoA ratio. | Up to 12 weeks
  The percentage change in liver injury and lipid metabolic indicators compared to the baseline period.
Hypersensitive C-reactive protein | Up to 12 weeks
  The change of hypersensitive C-reactive protein from baseline.
MRI-PDFF relative baseline decrease percentage | Baseline to Day 85
  Percentage of participants with a relative decrease in fat content (%) assessed by MRI-PDFF of ≥30% compared to baseline.
ALT relative to baseline decrease ratio | Up to 12 weeks
  The proportion of participants whose ALT decreased by more than 17 U/L compared to the baseline.
Fasting blood glucose, fasting insulin level, HOMA-IR, HbA1c, body weight, and BMI. | Up to 12 weeks
  Changes in glucose metabolism related indicators compared to baseline.
Cmax | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: Maximum observed plasma concentration.
Tmax | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: time to the maximum observed plasma concentration.
T1/2 | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: elimination half-life.
CL/F | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: apparent total plasma clearance.
Vd/F | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: apparent volume of distribution.
AUC0-∞ | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: AUC from time zero to infinity.
AUC0-24h | Up to 12 weeks
  Single-Dose Pharmacokinetic (PK) Parameter: AUC from time zero to 24 hours.
Cmax,ss | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: Steady-state peak concentration.
Tmax,ss | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: steady-state time to peak.
Cmin,ss | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: steady-state trough concentration.
Cavg,ss | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: mean steady-state blood drug concentration.
T1/2,ss | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: elimination half-life.
AUCtau | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: AUC over one dosing interval.
Rac | Up to 12 weeks
  Multiple-Dose Pharmacokinetic (PK) Parameter: accumulation factor.
The percentage change of sex hormone-binding globulin (SHBG) from baseline. | Up to 12 weeks
  Pharmacodynamics
Change in the Health Survey Short Form (SF-36) relative to baseline. | Baseline to day 85
  Patient-reported outcome

OTHER OUTCOMES:
Use iLivTouch to evaluate the changes of Liver stiffness measurement value (LSM) and Ultrasonic attenuation parameter (UAP) compared to the baseline. | Day 1, day 85.
  The influence of CS060380 tablets on improving fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Junping Shi, MD, Principal Investigator — The Affiliated Hospital of Hangzhou Normal University
Locations (4):
- China (4):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang